CLINICAL TRIAL: NCT04597554
Title: Influence of 8-Weeks Cranberry Supplementation on the Antibody Response to Influenza Vaccination and Ex-Vivo Viral Defense
Brief Title: Cranberry Supplementation, Viral Defense, Antibody Response to the Flu Shot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-0301
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Nutrition Immunology
Keywords: cranberry; influenza vaccination; antibody; viral defense
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry (Experimental): 4 oz. cranberry beverage (breakfast) and 2 chewable cranberry gummies (lunch) per day for 8 weeks.
  Interventions: Dietary Supplement: Cranberry
- Placebo (Placebo Comparator): 4 oz. placebo beverage (breakfast) and 2 chewable placebo gummies (lunch) per day for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry — Cranberry beverage and gummies supplement
  Arms: Cranberry
Dietary Supplement: Placebo — Placebo beverages and gummies supplement
  Arms: Placebo

SUMMARY:
This study will investigate the effect of 8-weeks cranberry supplementation on the antibody response to influenza vaccination and ex-vivo anti-viral activity. The hypothesis is that 8-weeks ingestion of cranberry supplement relative to placebo will improve the antibody response to influenza vaccination and ex-vivo anti-viral defense.

DETAILED DESCRIPTION:
Participants (n=90, ages 40-80 y) will be randomized to cranberry or placebo groups (with groups balanced for age, BMI, sex). Participants will provide blood and urine samples (lab visit #1), ingest cranberry or placebo supplements for 4-weeks, provide blood and urine samples and be vaccinated for influenza (lab visit #2), and provide two additional blood and urine samples after 1- (lab visit #3) and 4- additional weeks of supplementation (lab visit #4). Blood samples will be tested for seroconversion rates and haemagglutination inhibition [HI] titres, and anti-viral activity against viral infected Hela cells.

Lab Visit #1, Pre-Study: Orientation and review of the consent form (with next morning follow-up visit to turn in the 24-h urine sample). 10-15 minutes The informed consent form, Medical Health Questionnaire (MHQ), and 1-week retrospective symptom log (SYMPLOG) will be sent to the subject via email prior to Lab Visit #1. The research staff under the direction of the Research Manager will call each participant, review research procedures and the consent form, and set up appointment times for Lab Visit #1. Participants will be told that they will sign the consent form during Lab Visit #1. Participants will report to the NCRC Human Performance Lab in Kannapolis in an overnight fasted state (no food or beverages other the water for 8 or more hours). The study manager will make a final review of the consent form with the study participant prior to obtaining voluntary consent. Once voluntary consent has been provided by the study participant, the completed Medical Health Questionnaire (MHQ) and 1-week retrospective symptom log (SYMPLOG) will be turned in. The MHQ includes questions on lifestyle and medical histories. The SYMPLOG includes questions on digestive health (constipation, heartburn, bloating, diarrhea, and nausea), hunger levels (morning, afternoon, and evening), energy levels (morning, afternoon, and evening), sickness (fever, cough, sore throat, stuffy nose, runny nose, and headache), pain (joint, muscle, and back), allergies, stress level, focus/concentration, and overall well-being. Participants will indicate responses using a 12-point Likert scale with 1 relating to "none at all", 6 "moderate", and 12 "very high". Height, weight, and body composition will be obtained (in a screened off area of the lab to ensure privacy) using the seca Medical Body Composition Analyzer 514 bioelectrical impedance scale (Hanover, MD). Blood samples will be taken from an antecubital vein with subjects in the seated position. Supplements for the first 4 weeks of the study will be provided. During visit #1, participants will be given a 3-day food record with thorough written and oral instructions on recording procedures (with food models). The 3-day food record will be completed on a Thursday, Friday, and Saturday sequence prior to visit #2. During visit #1, participants will be given two 24-h urine collection kits with thorough written and oral instruction on collection procedures. The first 24-h urine collection bottles will be collected during the 24-h period immediately after lab visit #1 and turned in the next morning. (To minimize contact, participants will stay in their cars and hand urine samples to a research staff member). Supplementation will start the day after lab visit #1. The second 24-h urine collection bottle will be collected during the 24-h period immediately prior to lab visit #2.

Lab Visit #2, 4-Week Time Point: Provide blood and urine samples and be vaccinated for influenza (10 to 15 min) Participants will report to the NCRC Human Performance Lab in Kannapolis after 4-weeks supplementation in an overnight fasted state (no food or beverages other the water for 8 or more hours). Participants will turn in the 3-day food record and the 24-h urine sample. Compliance to the supplementation regimen will be reviewed and subjects will be asked to return all unused supplements. Participants will fill in the 1-week retrospective symptom log (SYMPLOG) before coming to the lab and turn in. Height, weight, and body composition will be obtained (in a screened off area of the lab to ensure privacy) using the seca Medical Body Composition Analyzer 514 bioelectrical impedance scale (Hanover, MD). Blood samples will be taken from an antecubital vein with subjects in the seated position.

Participants will receive the influenza vaccination for the 2020-21 season (in accordance with the CDC's Advisory Committee on Immunization Practices regarding the use of seasonal influenza vaccines in the United States). The influenza vaccination will not be administered by this study. The vaccinations will be provided by Walgreens personnel at the NCRC using standard procedures. Participants will receive the flu shot as clinically indicated by their physician or personnel administering the vaccine. The determination that the flu shot is not clinically indicated will also be determined by the participant's physician or personnel administering the vaccine. The high-dose vaccine will be used for study participants aged 65 years and older. (Note: Walgreens has provided influenza vaccinations at the NCRC for several years and have consented to provide them for our study participants. Participants will complete standard forms and present their insurance cards to cover the fee).

Supplements for the final 4 weeks of the study (weeks 5 through 8) will be provided. Participants will be given two 24-h urine collection bottles for Lab Visits #3 and #4.

Lab Visit #3, 5-Week Time Point: Provide blood and urine samples (10 min) Participants will report to the NCRC Human Performance Lab in Kannapolis at the 5-week time point in an overnight fasted state (no food or beverages other the water for 8 or more hours). Participants will turn in the 24-h urine sample. Compliance to the supplementation regimen will be reviewed and subjects will be asked to return all unused cranberry/placebo supplements. Participants will fill in the 1-week retrospective symptom log (SYMPLOG) before coming to the lab and turn in. Height, weight, and body composition will be obtained (in a screened off area of the lab to ensure privacy) using the seca Medical Body Composition Analyzer 514 bioelectrical impedance scale (Hanover, MD). Participants will remove their shoes and socks for the seca BIA measurement while holding the side rails. Blood samples will be taken from an antecubital vein with subjects in the seated position.

Lab Visit #4, 8-Week Time Point (end of study): Provide final blood and urine samples (10 min) Participants will report to the NCRC Human Performance Lab in Kannapolis at the 8-week time point in an overnight fasted state (no food or beverages other the water for 8 or more hours). Participants will turn in the 24-h urine sample. Compliance to the supplementation regimen will be reviewed. Participants will fill in the 1-week retrospective symptom log (SYMPLOG) before coming to the lab and turn in. Height, weight, and body composition will be obtained (in a screened off area of the lab to ensure privacy) using the seca Medical Body Composition Analyzer 514 bioelectrical impedance scale (Hanover, MD). Blood samples will be taken from an antecubital vein with subjects in the seated position.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written Informed Consent and follow verbal and written study directions in English.
* Adult men and women between ages 40-80 years.
* Body Mass Index (BMI) 25 to 40 kg/m2 (overweight, mild and moderate obesity).
* Must not be taking or be willing to stop taking cranberries or any products and supplements containing cranberries for seven days prior to the start of the study and for the duration of the study.
* Must not be taking or be willing to stop taking supplements containing probiotics, or polyphenols and flavonoids (e.g., quercetin, anthocyanins, green tea extract) for seven days prior to the start of the study and for the duration of the study.
* Able to maintain consistent diet and lifestyle habits throughout the study.
* Healthy, noninstitutionalized participants or those with chronic but stable and well controlled medical conditions (i.e., hypertension controlled by a consistent dose of medication for a minimum of six months; chronic use of consistent dose of blood-thinning medication; diet-controlled Type II diabetes; statin controlled high blood cholesterol) may participate at the discretion of the primary investigator (PI).
* Willing and able to provide fasting blood samples and 24-hour urine samples.
* Able to attend four scheduled visits at the AppState Human Performance Laboratory at the North Carolina Research Campus facility in Kannapolis, NC.
* Willing to receive the 2020-21 seasonal influenza vaccination (with high-dose vaccinations given to those 65 years of age and older, as recommended by the Centers for Disease Control and Prevention).

Exclusion Criteria:

* Current active treatment for heart disease or cancer (excluding skin cancer), or medically complicated conditions (i.e., diabetes requiring insulin, uncontrolled high blood pressure), at the discretion of the primary investigator.
* Inability to provide a venous blood sample or 24-hour urine sample.
* Unable or unwilling to provide written informed consent for participation in study.
* History of allergic reactions to cranberry juice or products containing cranberries.
* Have already received the 2020-21 seasonal influenza vaccination.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Serum IgG and IgG1 | Change from pre-study to 1 and 4 weeks post-flu shot (at the 4-week time point)
  Serum concentrations for IgG and IgG1 for the 3 specific influenza vaccine strains

SECONDARY OUTCOMES:
Anti-Viral Activity | Change from pre-study to post-supplementation after 4, 5, and 8 weeks
  Serum antiviral activity and viral replication using the vesicular stomatitis virus

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Upon request; de-identified data